CLINICAL TRIAL: NCT06267911
Title: Efficacy and Safety of a Non-immersive Virtual Reality-based Neuropsychological Intervention for Cognitive Stimulation and Psychological Support of Critical Care Patients
Brief Title: Rehabilitation Gaming System for Intensive Care Units
Acronym: RGS-ICU
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Collaborators: Corporacion Parc Tauli (Other); Hospital Son Llatzer (Other); Fundació La Marató de TV3 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202223-10; 160/U/2022 (Other Grant/Funding Number: Fundació La Marató de TV3)
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive stimulation and psychological support (RGS-ICU) (Experimental)
  Interventions: Other: Cognitive stimulation and psychological support (RGS-ICU)
- Treatment as usual (TAU) (No Intervention)

INTERVENTIONS:
Other: Cognitive stimulation and psychological support (RGS-ICU) — The RGS-ICU intervention consists of daily 20-minute sessions of early cognitive stimulation and psychological support adjuvant to standard ICU care administered by research staff and supervised by clinical staff each morning in the patient's own room during ICU admission and until ICU discharge or up to a maximum of 28 days after randomization. The sessions consist of orienting the patient to space and time, cognitive training of attention, working memory, learning/memory, executive function and processing speed, viewing of relaxing videos inspired by nature and fantasy scenarios to reduce stress and anxiety, and psychoeducation about the ICU environment and the characteristics of the cognitive, mental and physical state of critically ill patients.
  Arms: Cognitive stimulation and psychological support (RGS-ICU)

SUMMARY:
Admission to an Intensive Care Unit (ICU) is a potentially traumatic experience for a mentally vulnerable person. Beyond the stress and anxiety associated with the ICU environment and medical procedures, survivors of critical illness are at risk of developing cognitive and psychological sequelae related to Post-Intensive Care Syndrome (PICS). These disorders are associated with high economic, medical and personal costs.

This trial aims to evaluate the efficacy of an innovative neuropsychological e-health intervention for early cognitive stimulation and psychological support of people in critical care, i.e. the Rehabilitation Gaming System for Intensive Care Units (RGS-ICU) intervention, in improving comfort during ICU admission and cognition and mental health three and 12 months after ICU discharge. The RGS-ICU intervention, applied as an adjunct to standard ICU care, is based on non-immersive virtual reality techniques and has been specifically designed and developed to suit the needs of people in critical care and the characteristics of the ICU environment. To ensure the safety of the intervention, participants' physiological parameters will be automatically recorded by advanced continuous monitoring systems as part of standard ICU care.

The investigators hypothesize that the cognitive stimulation and psychological support protocols of the RGS-ICU intervention, applied as an adjunct to standard ICU care, in addition to being safe for people in critical care units, will improve comfort during ICU admission and cognitive and mental health outcomes after ICU discharge, compared to receiving standard ICU care alone.

The findings derived from this trial may contribute to establish a novel and superior paradigm of human-centered ICU care to improve the comfort of people admitted to the ICU. This achievement could also have a relevant impact on medical and economic costs during ICU admission, and on functionality and health-related quality of life after ICU discharge associated with the reduction of cognitive and psychological sequelae linked to PICS.

The RGS-ICU intervention has been designed at Corporacion Parc Taulí with the collaboration of the University of the Balearic Islands and has been developed by Eodyne Systems S.L., a company dedicated to the development of science-based technological solutions for intervention, monitoring, diagnosis, and prognosis in stroke and other brain disorders.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years)
* Admitted to a medical/surgical ICU
* For respiratory failure, cardiogenic shock, or septic shock
* With an expected ICU stay of ≥48 hours
* Residing in Catalonia or Majorca (Balearic Islands)
* Who speak Catalan and/or Spanish
* Who are able to give informed consent by themselves or through an authorized representative

Exclusion Criteria:

* History of intellectual disability or other neurodevelopmental disorders, such as autism spectrum disorder
* History of neurological disorders, dementia or other neurodegenerative diseases, such as epilepsy, Alzheimer's disease, Parkinson's disease or multiple sclerosis
* History of brain damage, such as traumatic brain injury or stroke
* History of severe psychiatric illness, such as psychotic, bipolar, depressive, obsessive-compulsive, post-traumatic or personality disorder
* Suspected or confirmed substance use disorder
* Suspected or confirmed communicable disease in an isolated patient
* Uncorrected hearing or visual impairment
* Any medical condition that prevents safe upper extremity mobility, such as skin lesions, burns, or fractures
* Life expectancy <12 months
* Enrolled in another trial that does not allow co-enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Attention performance | 12 months after discharge from the ICU
  Difference in attention performance (Z scores) between experimental and non-intervention groups assessed with the Wechsler Adult Intelligence Scale-IV (WAIS-IV) Forward Digit Span subtest 12 months after ICU discharge. Z scores have a mean of 0 and a standard deviation of 1. Higher scores indicate better attention performance.
Working memory performance | 12 months after discharge from the ICU
  Difference in working memory performance (Z scores) between experimental and non-intervention groups assessed with the WAIS-IV Backward Digit Span subtest 12 months after ICU discharge. Z scores have a mean of 0 and a standard deviation of 1. Higher scores indicate better working memory performance.
Learning/memory performance | 12 months after discharge from the ICU
  Difference in learning/memory performance (Z scores) between experimental and non-intervention groups assessed with the Rey Auditory Verbal Learning Test (RAVLT) 12 months after ICU discharge. Z scores have a mean of 0 and a standard deviation of 1. Higher scores indicate better learning/memory performance.
Executive function performance | 12 months after discharge from the ICU
  Difference in executive function performance (Z scores) between experimental and non-intervention groups assessed with the Trail Making Test (TMT), the Stroop Color and Word Test (SCWT), and the verbal phonemic fluency (FAS) test 12 months after ICU discharge. Z scores have a mean of 0 and a standard deviation of 1. Higher scores indicate better executive function performance.
Processing speed performance | 12 months after discharge from the ICU
  Difference in processing speed performance (Z scores) between experimental and non-intervention groups assessed with the WAIS-IV Digit Symbol-Coding subtest and the Symbol Digit Modalities Test (SDMT) 12 months after ICU discharge. Z scores have a mean of 0 and a standard deviation of 1. Higher scores indicate better executive function performance.
Incidence of Treatment-Emergent Adverse Events [Safety] | From ICU admission to ICU discharge or up to a maximum of 28 days after randomization
  Number of interrupted sessions due to adverse events in the patients' physiological parameters (oxygen saturation, respiratory rate and heart rate) during admission to the ICU. The higher the number of interrupted sessions, the less safe the intervention.

SECONDARY OUTCOMES:
Dyspnea intensity | From ICU admission to ICU discharge or up to a maximum of 28 days after randomization
  Change in dyspnea intensity before and after the intervention evaluated with a Visual Analogue Scale (VAS) with range 0-10. Higher scores indicate more intense dyspnea.
Pain intensity | From ICU admission to ICU discharge or up to a maximum of 28 days after randomization
  Change in pain intensity before and after the intervention evaluated with a Visual Analogue Scale (VAS) with range 0-10. Higher scores indicate more intense pain.
Worry intensity | From ICU admission to ICU discharge or up to a maximum of 28 days after randomization
  Change in worry intensity before and after the intervention evaluated with a Visual Analogue Scale (VAS) with range 0-10. Higher scores indicate more intense worry.
Sadness intensity | From ICU admission to ICU discharge or up to a maximum of 28 days after randomization
  Change in sadness intensity before and after the intervention evaluated with a Visual Analogue Scale (VAS) with range 0-10. Higher scores indicate more intense sadness.
Comfort experienced | Discharge from the ICU
  Difference in experienced comfort between experimental and non-intervention groups assessed with the Patient Evaluation of Emotional Comfort Experienced (PEECE) questionnaire at ICU discharge, a 12-item instrument with range 0-48. Higher scores indicate better subjective psychological well-being.
Anxiety symptoms | 12 months after discharge from the ICU
  Difference in anxiety symptoms between experimental and non-intervention groups assessed with the Generalized Anxiety Disorder (GAD-7) questionnaire 12 months after ICU discharge, a 7-item instrument with range 0-21. Higher scores indicate more severe anxiety symptoms.
Symptoms of depression | 12 months after discharge from the ICU
  Difference in symptoms of depression between experimental and non-intervention groups assessed with the Patient Health Questionnaire-9 (PHQ-9) 12 months after ICU discharge, a 9-item instrument with range 0-27. Higher scores indicate more severe symptoms of depression.
Symptoms of post-traumatic stress disorder | 12 months after discharge from the ICU
  Difference in post-traumatic stress disorder symptoms between experimental and non-intervention groups assessed with the Treatment-Outcome Post-Traumatic Stress Disorder Scale (TOP-8) 12 months after ICU discharge, a 8-item instrument with range 0-32. Higher scores indicate more severe symptoms of post-traumatic stress disorder.

OTHER OUTCOMES:
Objective cognition | 12 months after discharge from the ICU
  Difference in objective cognition between experimental and non-intervention groups assessed with the Montreal Cognitive Assessment (MoCA) 12 months after ICU discharge, a screening instrument with range 0-30. Higher scores indicate better objective cognitive performance.
Subjective cognition | 12 months after discharge from the ICU
  Difference in subjective cognition between experimental and non-intervention groups assessed with the Perceived Deficits Questionaire-5 (PDQ-5) 12 months after ICU discharge, a 5-item instrument with range 0-20. Higher scores indicate greater perceived cognitive deficits.
Functionality | 12 months after discharge from the ICU
  Difference in functionality between experimental and non-intervention groups assessed with the self-reported 12-item version of the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) 12 months after ICU discharge, an instrument with range 0-100. Higher scores indicate worse functionality.
Health-related quality of life | 12 months after discharge from the ICU
  Difference in health-related quality of life between experimental and non-intervention groups assessed with the 12-item Short-Form Health Survey (SF-12) 12 months after ICU discharge, an instrument with range 0-100. Higher scores indicate better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Navarra-Ventura, PhD, Principal Investigator — University of the Balearic Islands
Locations (3):
- Spain (3):
  - University of the Balearic Islands, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Son Llàtzer, Palma de Mallorca, Balearic Islands
  - Corporacion Parc Tauli, Sabadell, Catalonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Godoy-Gonzalez M, Lopez-Aguilar J, Fernandez-Gonzalo S, Goma G, Blanch L, Brandi S, Ramirez S, Blasi J, Verschure P, Rialp G, Roca M, Gili M, Jodar M, Navarra-Ventura G. Efficacy and safety of a non-immersive virtual reality-based neuropsychological intervention for cognitive stimulation and relaxation in patients with critical illness: study protocol of a randomized clinical trial (RGS-ICU). BMC Psychiatry. 2024 Dec 18;24(1):917. doi: 10.1186/s12888-024-06360-4. PMID 39696098